CLINICAL TRIAL: NCT02757781
Title: Effectiveness of a Virtual Intervention (CoP) for Professionals to Improve Their Attitude Towards the Empowerment of Patients With Chronic Disease: Cluster Randomised Controlled Trial (eMPODERA Project)
Brief Title: Effectiveness of a Virtual Intervention for Professionals to Improve Their Attitudes Towards Patient Empowerment.
Acronym: eMPODERA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Avedis Donabedian Research Institute (Other)
Collaborators: Servicio Canario de Salud (Other); Gerencia de Atención Primaria, Madrid (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PI15/00164
Record Dates: First submitted 2016-04-25; First posted 2016-05-02 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Disease
Keywords: Patient empowerment; Patient involvement; Patient participation; Healthcare professional attitudes; Chronic diseases
MeSH Terms: conditions — Chronic Disease; Patient Participation | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Group of healthcare professionals that NOT receive the intervention (community of practice)
- Intervention group (Experimental): Group of healthcare professionals that receive the intervention (community of practice)
  Interventions: Behavioral: Community of Practice

INTERVENTIONS:
Behavioral: Community of Practice — The intervention group will be offered participation for 12 months in a virtual CdP based on a web 2.0 platform. The control group will receive usual training.
  Other Names: educational intervention
  Arms: Intervention group

SUMMARY:
The eMPODERA study aims to assess the effectiveness of a Community of Practice (CdP) virtual in improving attitudes of primary care professionals on the empowerment of patients with chronic diseases.

DETAILED DESCRIPTION:
Main Objective: to assess the effectiveness of a Community of Practice (CdP) virtual in improving attitudes of health professionals in primary care on the empowerment of patients with chronic diseases.

Methodology:

Design: cluster randomised controlled.

Scope: primary care centers (PCC) belonging to the Regions of Catalonia, Madrid and Canary Islands.

Population: primary care health professionals (family doctors and nurses).

Sample size: 270 healthcare professionals and 1382 patients.

Randomization: Randomization unit: PCC; unit of analysis: primary care health professionals. 9 pairs of PCC by region will be randomly selected and randomly assigned to the intervention or control group. Randomization will be performed after the selection of professionals and patients.

Intervention: the intervention group will be offered participation for 12 months in a virtual CdP based on a web 2.0 platform. The control group will receive usual training.

Measurements: the primary outcome will be measured by Patient-Provider Orientation Scale (PPOS) questionnaire at baseline and 12 months. Secondary outcomes: sociodemographic of professionals; sociodemographic and clinical characteristics of patients; Patient Activation Measure (PAM) questionnaire for patient activation; outcomes regarding use of the CdP.

Analysis: A linear mixed-effects regression to estimate the effect of participating in the CdP will be estimated. Additionally, an analysis of how the CdP is functioning through techniques of social network analysis and control charts will be performed.

ELIGIBILITY:
Inclusion Criteria:

Clusters:

* Primary Care Centres (PCC) with Electronic Record system with more than 1 year of implementation
* PCC belongs to the Automonous Comunities of Canary Island, Catalonia and Madrid

Healthcare professionals:

* Acceptance to participate
* stable contract with the Primary care centre
* Physician or Nurses

Exclusion Criteria:

Clusters:

- Primary Care Centres where its directors do not accept to participate in the trial

Healthcare professionals:

* Students
* Medical and Nursing residents

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from Patient-Provider Orientation Scale (PPOS) at 12 months | At baseline and 12 months
  PPOS is a questionnaire administrated to healthcare professionals

SECONDARY OUTCOMES:
Change from Patient Activation Measure (PAM) at 12 months | Baseline and 12 months
  PAM is validated questionnaire to measure patient activation (administrated to patients)

CONTACTS AND LOCATIONS:
Overall Officials: Carola Orrego, PhD, Principal Investigator — Avedis Donabedian Research Institute; Lilisbeth Perestelo, PhD, Principal Investigator — Servicio de Evaluación del Servicio Canario de la Salud; Ana I Gonzalez, MD, Principal Investigator — Unidad de Apoyo Técnico de la Gerencia Asistencial de Atención Primaria de la Comunidad de Madrid; Carlos Bermejo, RN,Msc, Principal Investigator — Unidad de Apoyo Técnico de la Gerencia Asistencial de Atención Primaria de la Comunidad de Madrid

IPD SHARING:
Plan to Share IPD: No
There is not plan to make individual participant data available

REFERENCES:
- [Derived] Koatz D, Torres-Castano A, Salrach-Arnau C, Perestelo-Perez L, Ramos-Garcia V, Gonzalez-Gonzalez AI, Pacheco-Huergo V, Toledo-Chavarri A, Gonzalez-Pacheco H, Orrego C. Exploring value creation in a virtual community of practice: a framework analysis for knowledge and skills development among primary care professionals. BMC Med Educ. 2024 Feb 7;24(1):121. doi: 10.1186/s12909-024-05061-6. PMID 38326814
- [Derived] Orrego C, Perestelo-Perez L, Gonzalez-Gonzalez AI, Ballester-Santiago M, Koatz D, Pacheco-Huergo V, Rivero-Santana A, Ramos-Garcia V, Fernandez NM, Torres-Castano A, Bermejo-Caja C. A Virtual Community of Practice to Improve Primary Health Care Professionals' Attitudes Toward Patient Empowerment (e-MPODERA): A Cluster Randomized Trial. Ann Fam Med. 2022 May-Jun;20(3):204-210. doi: 10.1370/afm.2799. PMID 35606139
- [Derived] Bermejo-Caja CJ, Koatz D, Orrego C, Perestelo-Perez L, Gonzalez-Gonzalez AI, Ballester M, Pacheco-Huergo V, Del Rey-Granado Y, Munoz-Balsa M, Ramirez-Puerta AB, Canellas-Criado Y, Perez-Rivas FJ, Toledo-Chavarri A, Martinez-Marcos M; e-MPODERA group. Acceptability and feasibility of a virtual community of practice to primary care professionals regarding patient empowerment: a qualitative pilot study. BMC Health Serv Res. 2019 Jun 20;19(1):403. doi: 10.1186/s12913-019-4185-z. PMID 31221215
- [Derived] Gonzalez-Gonzalez AI, Orrego C, Perestelo-Perez L, Bermejo-Caja CJ, Mora N, Koatz D, Ballester M, Del Pino T, Perez-Ramos J, Toledo-Chavarri A, Robles N, Perez-Rivas FJ, Ramirez-Puerta AB, Canellas-Criado Y, Del Rey-Granado Y, Munoz-Balsa MJ, Becerril-Rojas B, Rodriguez-Morales D, Sanchez-Perruca L, Vazquez JR, Aguirre A. Effectiveness of a virtual intervention for primary healthcare professionals aimed at improving attitudes towards the empowerment of patients with chronic diseases: study protocol for a cluster randomized controlled trial (e-MPODERA project). Trials. 2017 Oct 30;18(1):505. doi: 10.1186/s13063-017-2232-9. PMID 29084597